CLINICAL TRIAL: NCT01372033
Title: Effects of Manualized Treatment in a Seamless System of Care: Handling Probation
Brief Title: Effects of Manualized Treatment in a Seamless System
Acronym: Man Tx
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: George Mason University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Faye S Taxman, Ph.D., Univeristy Professor, George Mason University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01DA017729 (NIH); R01DA017729 (NIH)
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2009-06

CONDITIONS: Substance Abuse; Offenders; Criminal Thinking; HIV Risk Behaviors
Keywords: drug treatment; substance abuse; offenders; high risk
MeSH Terms: conditions — Substance-Related Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CBT (Experimental): Use of cognitive behavioral therapy focused on social skill development and interpersonal relationships
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 18 sessions of CBT, twice weekly
Behavioral: Cognitive Behavioral Therapy — 18 sessions with goals groups drug testing

SUMMARY:
The specific aims of this project are:

1. To conduct a randomized block experiment to test the effectiveness of different models of the seamless supervision/treatment system and traditional criminal justice supervision on reducing recidivism and drug use, and improving social adjustment among offenders;
2. To understand the differential impacts based on offender risk factors (e.g., propensity to engage in further criminal behavior) on criminal justice outcomes and to determine whether differences found between seamless and traditional system participants are moderated by offender risk level;
3. To understand differential treatment and social adjustment outcomes (e.g., treatment progress, employment status) of different types of offenders participating in various treatment services; and
4. To examine levels of systems and service integration between the supervision and treatment systems pre- and post-intervention and to measure the impact of integration on outcomes over time.

ELIGIBILITY:
Inclusion Criteria:

* Substance abusers

  * men and women
  * treatment

Exclusion Criteria:

* Parolees

  * Low threshold substance abuse
  * violent offenders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2007-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Arrest | 12 months

SECONDARY OUTCOMES:
Treatment Completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Faye S Taxman, Ph.D., Principal Investigator — George Mason University
Locations (1):
- Maryland Dvision of Parole and Probation, Baltimore, Maryland, United States